CLINICAL TRIAL: NCT06500299
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Safety and Efficacy of HDM1002 Tablets in Overweight and Obese Adults
Brief Title: Evaluate the Safety and Efficacy of HDM1002 Tablets in Overweight and Obese Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM1002-201
Record Dates: First submitted 2024-06-13; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity
Keywords: HDM1002 tablet; overweight and obesity; Glucagon-Like Peptide-1 Receptor Agonists
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HDM1002 100mg BID (Experimental): HDM1002 tablets 100mg twice daily, 12weeks
  Interventions: Drug: HDM1002 100 mg QD
- HDM1002 200mg BID (Experimental): HDM1002 tablets 200mg twice daily, 12weeks
  Interventions: Drug: HDM1002 200 mg QD 12weeks
- HDM1002 400mg QD (Experimental): HDM1002 tablets 400mg once daily, 12weeks
  Interventions: Drug: HDM1002 400 mg QD 12weeks
- placebo (Placebo Comparator): Matching placebo will be provided， 12weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HDM1002 100 mg QD — HDM1002 tablets 100mg daily, 12weeks
  Other Names: HDM1002
  Arms: HDM1002 100mg BID
Drug: HDM1002 200 mg QD 12weeks — HDM1002 tablets 200mg daily, 12weeks
  Other Names: HDM1002
  Arms: HDM1002 200mg BID
Drug: HDM1002 400 mg QD 12weeks — HDM1002 tablets 400mg daily, 12weeks
  Other Names: HDM1002
  Arms: HDM1002 400mg QD
Drug: Placebo — Matching placebo will be provided
  Arms: placebo

SUMMARY:
It is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the safety and efficacy of HDM1002 tablets in overweight and obese adults.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled phase II clinical trial aims to evaluate the safety and efficacy of HDM1002 tablets in overweight and obese adults. Participants with a BMI between 24 and 40 will be include. A total of 180 participants will be randomized in a 1:1:1:1 ratio to receive different doses of HDM1002 or placebo. Following the screening period to confirm eligibility up to 2-weeks, the study will consist of a treatment period will be 12 weeks, followed by an approximate 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age (inclusive).
* BMI≥28 but < 40.0 kg/m2 at screening or randomization，or BMI≥24.0 kg/m2 but < 28 kg/m2 with any of the following:

  1. Hypertension
  2. Impaired fasting glucose or impaired glucose tolerance
  3. Dyslipidemia
  4. Obstructive sleep apnea syndrome
* At least one previous failure to lose weight through lifestyle modification was defined as < 5% weight loss after ≥3 months of lifestyle modification.

Exclusion Criteria:

* Weight change ≥5% as reported or documented. Previous diagnosis of type 1, type 2, or any other type of diabetes.
* Diagnosis of overweight or obesity due to other diseases or medications.
* History or family history of medullary thyroid carcinoma, C cell hyperplasia, or multiple endocrine neoplasia type 2.
* Have diseases or conditions that affect gastric emptying or gastrointestinal absorption of nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, chronic pancreatitis, etc. Or a history of acute pancreatitis or acute gallbladder disease within 3 months before signing ICF.
* GLP-1R agonist use within 6 months prior to signing ICF.
* Use of hypoglycemic drugs within 3 months before signing ICF.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change From Baseline in Body Weight at Week 12 | Baseline, Week 12
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Percentage Change From Baseline in Body Weight at Week 2, Week 4, Week 6, Week 8, Week 10 | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg.
Percentage Change of Participants Achieving Weight Loss ≥ 5% and ≥ 10% at Week 12 | Baseline, Week 12
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg.
Change From Baseline in Body Mass Index (BMI), And Waist Circumference | Baseline, Week 12
  BMI was recorded in kg/m2, and Waist Circumference was recorded in cm
Percentage change from baseline in fasting lipid profile (total cholesterol, low density lipoprotein [LDL] cholesterol, high density lipoprotein [HDL] cholesterol, non HDL cholesterol, lipoprotein (a) (Lp[a]), triglycerides) | Baseline, Week 12
  Fasting Lipid Profiles were measured at planned time points.
Change From Baseline in Systolic and Diastolic Blood Pressure | Baseline, Week 12
  Blood Pressure was measured using an automated device
Number of Participants with Clinical Laboratory Abnormalities, and Abnormalities in Vital Signs, Physical Examination and Electrocardiogram and Number of Participants With Treatment Emergent Adverse Events | Through Week 16]
  Vital signs (blood pressure, pulse rate, body temperature, respiratory rate), physical examination, ECG and clinical laboratory evaluations (hematology, clinical chemistry, coagulation, urinalysis, calcitonin, serum amylase and lipase)

OTHER OUTCOMES:
Change From Baseline in Fasting Insulin | Time Frame: Baseline, Week 12
  The fasting plasma glucose measures the levels of Fasting Insulin were measured at planned time points
Change From Baseline in Fasting plasma Glucose | Time Frame: Baseline, Week 12
  The fasting plasma glucose measures the levels of glucose in the bloodFasting Insulin were measured at planned time points
Change From Baseline in Fasting C-Peptide, | Time Frame: Baseline, Week 12
  The fasting plasma glucose measures the levels of C-Peptide were measured at planned time points
Change From Baseline in HbA1c at Week 12 | Time Frame: Baseline, Week 12
  HbA1c can be used as a diagnostic test for diabetes and is a widely recognized objective measure of glycemic control
Pharmacokinetic (PK) Profiles of HDM1002 and Its Metabolites (If Feasible) | Day 1, Day 15, Day 29, Day 57 and Day 85
  Area under the curve from time 0 to 24 h(AUC0-24h)
Pharmacokinetic (PK) Profiles of HDM1002 and Its Metabolites (If Feasible) | Day 1, Day 15, Day 29, Day 57 and Day 85
  Maximum plasma concentration (Cmax),
Pharmacokinetic (PK) Profiles of HDM1002 and Its Metabolites (If Feasible) | Day 1, Day 15, Day 29, Day 57 and Day 85
  Minumum plasma concentration (Cmin)
Pharmacokinetic (PK) Profiles of HDM1002 and Its Metabolites (If Feasible) | Day 1, Day 15, Day 29, Day 57 and Day 85
  Time to maximum plasma concentration (Tmax)
Pharmacokinetic (PK) Profiles of HDM1002 and Its Metabolites (If Feasible) | Day 1, Day 15, Day 29, Day 57 and Day 85
  AUCtau

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Principal Investigator — Zhongshan Hospital, Shanghai, China